CLINICAL TRIAL: NCT02766348
Title: Randomized, Controlled Study of the Safety and Efficacy of DC-CTL Immune Cell for Non-Small Cell Lung Cancer
Brief Title: Clinical Efficacy and Safety of Dendritic Cytotoxic Lymphocyte(DC-CTL) Cell Infusion in NSCLC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Hornetcorn Bio-technology Company, LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYK-DC-CTL-NSCLC
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: NSCLC
Keywords: DC-CTL, NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DC-CTL (Experimental): After accepting chemotherapy of gGemcitabine and Cisplatin according to National comprehensive Cancer Network(NCCN) guidelines, patients will receive 3 cycles of DC-CTL treatment
  Interventions: Drug: gemcitabine; Biological: DC-CTL; Drug: cisplatinum
- Chemotherapy (Active Comparator): After accepting chemotherapy of Gemcitabine and Cisplatin according to NCCN guidelines, patients will just regularly follow up.
  Interventions: Drug: gemcitabine; Drug: cisplatinum

INTERVENTIONS:
Drug: gemcitabine — gemcitabine 1000mg/m2 IV on day 1 an day 8, repeat every 3 weeks
  Other Names: Gemzar
Biological: DC-CTL — 8×10^9 DC-CTL cells for each infusion, IV(In the vein) for 3 cycles, each cycle received four infusions on day 14,16,30 and 32
  Arms: DC-CTL
Drug: cisplatinum — cisplatin 25mg/m2 IV on day 1,2 and 3, repeat every 3 weeks.

SUMMARY:
Patients in group A will receive DC-CTL treatment and chemotherapy. Patients in group B will receive only chemotherapy.

DETAILED DESCRIPTION:
60 patients with stage III-IV NSCLC will be randomly divided into group A (receive DC-CTL treatment with chemotherapy) or group B (Just receive chemotherapy), and the randomize ratio will be 1:1, patients in group A will receive 3 cycles of DC-CTL treatment (every 1 months) and 4 cycles of chemotherapy (every 2 weeks). Patients in group B will receive only 4 cycles chemotherapy(every 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* The patient who have signed the informed consent;
* Histologically confirmed with NSCLC at stage III-IV
* Expected survival time is more than 2 month;
* Eastern Cooperative Oncology Group(ECOG) performance status was 0-2

Exclusion Criteria:

* Hemoglobin <8.0 g/dL, White blood cell <3 x 10^9/L; Platelet count <75 x 10^9/L; alanine aminotransferase(ALT), aspartate aminotransferase(AST), blood urea nitrogen(BUN) and Creatinine(CR) more than normal limits on 3.0 times;
* Known or suspected allergy to the investigational agent or any agent given in association with this trial;
* Pregnant or lactating patients;
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV) or TreponemaPallidun (TP) infection;
* Patients who are suffering from serious autoimmune disease;
* Patients who had used long time or are using immunosuppressant;
* Patients who had active infection;
* Patients who are suffering from serious organ dysfunction;
* Patients who are suffering from other cancer;
* Other situations that the researchers considered unsuitable for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Zi L Zhang, researcher, Study Director — Jingzhou Central Hospital
Locations (1):
- Jingzhou Central hospital Immunotherapy center, Jingzhou, Hubei, China

IPD SHARING:
Plan to Share IPD: No